CLINICAL TRIAL: NCT03171727
Title: Post-TIPS Short-term Low Molecular Weight Heparin for the Prevention of Early TIPS Dysfunction
Brief Title: Low Molecular Weight Heparin for the Prevention of Early TIPS Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, attending doctor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMWH-TIPS
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Liver Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): After TIPS procedure was performed, low molecular weight heparin was given for three days.
  Interventions: Drug: low molecular weight heparin
- control group (No Intervention): After TIPS procedure was performed, no low molecular weight heparin was given.

INTERVENTIONS:
Drug: low molecular weight heparin — After TIPS procedure was performed, low molecular weight heparin was given for three days.
  Arms: study group

SUMMARY:
Transjugular intrahepatic portosystemic shunt (TIPS) dysfunction is defined as a loss of decompression of the portal venous system due to occlusion or stenosis of the TIPS. Occlusion of the TIPS can either be due to thrombosis or hyperplasia of the intima. Thrombosis of the TIPS usually occurs early and can happen within 24 hours of TIPS creation. The frequency of this complication is on the order of 10%-15% when bare stents are used. Post-TIPS short-term low molecular weight heparin (LMWH) was used to prevent the early thrombosis formation. Weather post-TIPS LMWH was necessary when polytetrafluoroethylene-covered stent was used during TIPS creation was not answered. The present study was designed to evaluate the effect of short-term use of LMWH on early TIPS dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of liver cirrhosis
2. Technical success of TIPS was achieved.

Exclusion Criteria:

1. Non-cirrhotic portal hypertension
2. Portal vein thrombosis
3. Budd-Chiari syndrome
4. Pregnancy
5. Contradictions to anticoagulation therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-05-15 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
TIPS patency rate | one year
  Analysis

SECONDARY OUTCOMES:
LMWH-related complication | one month
  Analysis
Mortality rate | one year
  Analysis

CONTACTS AND LOCATIONS:
Overall Officials: xuefeng luo, Principal Investigator — Sichuan University
Locations (1):
- West china Hospital, Chengdu, China

IPD SHARING:
Plan to Share IPD: Undecided